CLINICAL TRIAL: NCT01860443
Title: Telepsychiatry-Based Collaborative Program to Improve the Management of Adolescent Depression in Primary Care Clinics in the Araucanía Region, Chile: A Randomized Controlled Trial
Brief Title: Telepsychiatry to Improve the Management of Adolescent Depression in Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because there are enough data to present the conclusions
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Vania Martínez-Nahuel, Dr.med., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONIS SA12I1294
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: depression; adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telepsychiatry collaborative program (Experimental): * Online training on the diagnosis and management of adolescent depression for health professionals from primary care clinics participating in active branch.
  * Clinical management of depression by primary care professionals, according to algorithms based on the Clinical Guidelines of the Chilean Ministry of Health (MINSAL).
  * Supervision of primary care professionals through an internet site run by a team of specialists.
  * Telephone monitoring of patients by personnel trained on clinical progress, treatment adherence, and side effects (applicable for patients taking drugs).
  Interventions: Other: Telepsychiatry collaborative program
- Usual care (Active Comparator): * Online training on the diagnosis and management of adolescent depression for health professionals from primary care centers participating in active branch.
  * Clinical management of depression by primary care professionals, according to algorithms based on the Clinical Guidelines of the Chilean Ministry of Health (MINSAL).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Telepsychiatry collaborative program — The intervention includes:
  * Online training for the health staff
  * Medical and psychological treatment, as described in the AUGE Clinical Guidelines for Depression
  * Online supervision in a web platform by specialists
  * Telephone monitoring
  Arms: Telepsychiatry collaborative program
Other: Usual care — * Online training for the health staff
  * Medical and psychological treatment, as described in the AUGE Clinical Guidelines for Depression
  Arms: Usual care

SUMMARY:
Background: Depression is common in adolescents and it is associated with serious consequences. In Chile, primary care team has a leading role in the management of depression in adolescents. Nevertheless, the majority of primary care professionals report not feeling adequately prepared to take on this responsibility and having difficulties referring patients to specialists. This situation is particularity complex in regions far away from the central zone. Telepsychiatry is a potential solution to an equitable access to specialized clinical expertise.

Purpose: The purpose of this study is to determine whether a telepsychiatry-based collaborative program is effective to improve the management of depression in adolescents between 13 and 19 years of age in 16 primary care clinics in the Araucanía Region, Chile.

Study design: A cluster-randomized clinical trial will be carried out with 237 adolescents. The efficacy, adherence, and acceptability of the telepsychiatry-based collaborative program will be evaluated.

DETAILED DESCRIPTION:
General aim To carry out a randomized controlled trial to compare the efficacy of telepsychiatry intervention versus usual care to treat depression in adolescents in primary care clinics in the Araucanía Region, Chile.

Specific aims

1. To compare the level of depressive symptoms of adolescents suffering depression participating in a telepsychiatry program versus usual care in primary care clinics.
2. To compare the level of health-related quality of life (HRQoL) of adolescents suffering depression participating in a telepsychiatry program versus usual care in primary care clinics.
3. To compare adolescents' adherence with a telepsychiatry program versus usual care in primary care clinics.
4. To evaluate adolescents' satisfaction with a telepsychiatry program.
5. To evaluate health staff's satisfaction with a telepsychiatry program.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria of a depressive disorder according a structured interview (MINI-KID)

Exclusion Criteria:

* Psychotic symptoms
* Bipolar disorder
* Current substance and/or alcohol dependence
* Suicide risk that requires specialized treatment
* Current treatment with antidepressant and/or psychotherapy
* Low intellectual abilities

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Beck Depression Inventory (BDI) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in KIDSCREEN-27 | Baseline and 12 weeks
  Health-related quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vania Martínez-Nahuel, Dr.med., Principal Investigator — University of Chile
Locations (7):
- Chile (7):
  - CESFAM Alemania, CESFAM Huequén, CESFAM Piedra de Águila, Angol
  - CESFAM Dr. Cristóbal Sáenz Cerda, Lautaro
  - CESFAM Nueva Imperial, Nueva Imperial
  - Consultorio Pitrufquén, Pitrufquén
  - CESFAM Amanecer, CESFAM Labranza, CESFAM Pedro de Valdivia, CESFAM Pueblo Nuevo, CESFAM Santa Rosa, CESFAM Villa Alegre, Consultorio Miraflores, Temuco
  - Hospital de Vilcún, Vilcún
  - CESFAM Villarrica, Villarrica

REFERENCES:
- [Derived] Martinez V, Rojas G, Martinez P, Zitko P, Irarrazaval M, Luttges C, Araya R. Remote Collaborative Depression Care Program for Adolescents in Araucania Region, Chile: Randomized Controlled Trial. J Med Internet Res. 2018 Jan 31;20(1):e38. doi: 10.2196/jmir.8021. PMID 29386172